CLINICAL TRIAL: NCT00852813
Title: Tolerance and Prebiotic Activity of Arabinoxylan-Oligosaccharides in Healthy Subjects: a Randomized, Placebo-Controlled Cross-Over Study
Brief Title: Tolerance and Prebiotic Activity of Arabinoxylan-Oligosaccharides in Healthy Subjects
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: KU Leuven (Other)
Responsible Party: Kristin verbeke, Katholieke Universiteit Leuven
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: AXOS 002
Record Dates: First submitted 2009-02-26; First posted 2009-02-27 (Estimated); Last update posted 2009-02-27 (Estimated); Status verified 2009-02

CONDITIONS: Healthy
Keywords: tolerance; prebiotic; gastrointestinal effects

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Dietary Supplement: arabinoxylan-oligosaccharides (AXOS) — intake period: 3 weeks, 10 g/day

SUMMARY:
The purpose of the study is to evaluate the tolerance of a higher dose of arabinoxylan-oligosaccharides (AXOS) and their prebiotic activity in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* healthy
* 18-45 years
* regular eating pattern

Exclusion Criteria:

* gastrointestinal complaints
* antibiotic intake
* medication influencing gut transit or microbiota
* abdominal surgery
* pregnancy

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2007-10; Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Verbeke, PhD, Study Director — KU Leuven
Locations (1):
- Department of Gastrointestinal Research, Laboratory Digestion and Absorption, Leuven, Leuven, Belgium

REFERENCES:
- [Background] Cloetens L, De Preter V, Swennen K, Broekaert WF, Courtin CM, Delcour JA, Rutgeerts P, Verbeke K. Dose-response effect of arabinoxylooligosaccharides on gastrointestinal motility and on colonic bacterial metabolism in healthy volunteers. J Am Coll Nutr. 2008 Aug;27(4):512-8. doi: 10.1080/07315724.2008.10719733. PMID 18978172